CLINICAL TRIAL: NCT06622291
Title: Efficacy of Nitric Oxide Administration for Reducing the Risk of Acute Kidney Injury in Patients With Acute Type A Aortic Dissection: a Randomized Controlled Trial
Brief Title: Perioperative Nitric Oxide Prevents Acute Kidney Injury in Acute Type A Aortic Dissection Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, chenzheyuan, MD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-16-20240626; Z191100006619095 (Other Grant/Funding Number: Beijing Municipal Science & Technology Commission); 2025AZB6001 (Other Grant/Funding Number: Beijing Anzhen Hospital High Level Research Funding)
Record Dates: First submitted 2024-09-24; First posted 2024-10-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Kidney Injury; Nitrous Oxide; Acute Type A Aortic Dissection
Keywords: Acute Kidney Injury; Nitrous Oxide; Aortic Dissection; cardiopulmonary bypass
MeSH Terms: conditions — Acute Kidney Injury; Aortic Dissection | interventions — Nitric Oxide

STUDY DESIGN:
Intervention Model Description: Single-center prospective, randomized, placebo-controlled study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide (Experimental): Patients in this group receive treatment with exogenous nitric oxide (NO) via the CPB machine. After CPB, NO is administered through the inspiratory limb of the anesthetic or ventilator circuit and then via the mechanical ventilator in the ICU. Once patients are extubated, they will breathe NO through a facemask or nasal cannula. NO administration begins at the start of CPB and continues for 12 hours post-operation.
  Interventions: Drug: Nitric Oxide
- Usual care (Placebo Comparator): Patients in this group receive a sham treatment without the supply of nitric oxide during CPB and for 12 hours post-operation.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nitric Oxide — Exogenous nitric oxide is directly administered to the oxygenator in the cardiopulmonary bypass circuit at a concentration of 60 ppm. Nitric oxide is also directly administered to the ventilator at a concentration of 60 ppm for 12 hours post-operation.
  Arms: Nitric Oxide
Other: Placebo — This is the placebo group. The standard CPB protocol involves delivering an air-gas mixture to the cardiopulmonary bypass circuit during cardiac surgery and avoiding the use of nitric oxide within 12 hours after surgery.
  Arms: Usual care

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of exogenous nitric oxide therapy in reducing the occurrence of acute kidney injury in patients with acute type A aortic dissection. Additionally, it aims to assess the safety of exogenous nitric oxide therapy.

DETAILED DESCRIPTION:
The incidence of acute kidney injury following acute type A aortic dissection is significantly high, thereby exerting a substantial impact on patient prognosis. Nitric oxide, an endogenous gaseous molecule with potential therapeutic effects, has been investigated in clinical studies as a treatment for acute kidney injury following cardiac surgery. However, there is currently no clinical study exploring the application of nitric oxide in patients with acute type A aortic dissection. Therefore, this study aims to investigate whether exogenous nitric oxide therapy has renal protective effects and its mechanism.

This prospective randomized study is conducted at Beijing Anzhen Hospital in Beijing, China. A total of 106 adult patients with acute type A aortic dissection are enrolled in this study. The patients are randomly divided into two groups: the experimental group received NO combined with conventional treatment, and the control group is only given conventional treatment. In the experimental group, 60 ppm NO is administered during intraoperative CPB and continued until within 12 hours after surgery.

The primary endpoint is the incidence of acute kidney injury (AKI) within 48 hours after surgery. The secondary endpoints include AKI grade (KDIGO); urine volume during CPB, within 12 and 24 hours after surgery; blood flow grade, resistance index, and pulsatility index in renal ultrasound at ICU admission, 12 and 24 hours after surgery; SOFA score at 24 hours after surgery; VIS score at ICU admission, 12 and 24 hours after surgery; duration of mechanical ventilation, non-invasive ventilation, and high-flow oxygen therapy; length of ICU stay and hospital stay; renal adverse events within 90 days; volume of drainage from the pleural and pericardial cavities after surgery. Additionally, dosage of diuretics and recombinant human brain natriuretic peptide during surgery and within 48 hours after surgery; oxygenation index and near-renal infrared oxygen saturation; levels of free hemoglobin, methemoglobin, nitrite (NO2-) and the total of NO metabolites (NOt); neutrophil gelatinase-associated lipocalin concentration; levels of the neutrophils lymphocytes ratio (NLR), the platelet lymphocyte ratio (PLR), systemic inflammatory response index (SIRI), and systemic immune response index (SII) ; CVP and PEEP, the volume of transfusions with plasma and stored or autologous RBCs will also be measured in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent;
2. Participants must be over 18 years of age;
3. Participants should meet the diagnostic and treatment guidelines for thoracic aortic diseases jointly issued by ACC/AHA in 2022, have received clinical and radiological diagnosis of acute type A aortic dissection, and undergone surgical thoracotomy within two weeks after symptom onset.

Exclusion Criteria:

1. Missing baseline value or missing postoperative serum creatinine value (Scr);
2. Preoperative eGFR less than 30ml/min/1.73m2 or receive renal replacement therapy;
3. History of kidney disease, including glomerular diseases: acute glomerulonephritis, rapidly progressive glomerulonephritis, chronic glomerulonephritis, nephrotic syndrome, etc., secondary nephropathy: lupus nephritis, diabetic nephropathy, interstitial nephritis, renal tubular disease, chronic renal failure, renal replacement therapy, etc.;
4. Previous renal tumor, kidney transplantation, and other related surgery;
5. Patients with single kidney;
6. History of malignant tumor or received radiotherapy and chemotherapy;
7. Severe skeletal muscle disease and autoimmune disease;
8. Preoperative dissection rupture or hemodynamic instability (systolic blood pressure <90mmHg);
9. Life expectancy less than 90 days;
10. Pregnant and lactating women, patients with mental disorders;
11. With intravascular or extravascular hemolytic disease;
12. Have participated in other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury (AKI) | 48 hours
  Incidence of Acute Kidney injury. The presence of acute kidney injury (AKI) is assessed during 48 hours after surgery. AKI is defined as follows: an increase in serum creatinine ≥ 0.3 mg/dL (≥ 26.5 μM/L) during 48 hours after surgery; or an increase in serum creatinine by ≥ 1.5 times compared with the initial preoperative level for seven days after intervention; or urine output < 0.5 mL/kg/h for 6 hours during the first 48 h after surgery.

SECONDARY OUTCOMES:
AKI grade | 48 hours after surgery
  Grade I: an increase in serum creatinine ≥ 0.3 mg/dL (≥ 26.5 μM/L) during 48 hours after surgery; or an increase in serum creatinine by ≥ 1.5 times compared with the initial preoperative level for seven days after the intervention; or urine output < 0.5 mL/kg/h for 6 hours during the first 48 h after surgery. Grade II: an increase in serum creatinine by 2-2.9 times compared with the initial preoperative level for seven days after the intervention. Grade III: an increase in serum creatinine by ≥ 3 times compared with the initial preoperative level for seven days after the intervention; or an increase in serum creatinine ≥ 4.0 mg/dL (≥ 353.6 μM/L) during 48 hours after surgery; or start RRT.
Urine output | During CPB surgery, 12 and 24 hours after surgery
  Urine output values (mL/kg/h) are assessed during CPB and 24 hours after surgery.
Vasoactive-inotropic score | immediate admission to ICU, 12 and 24 hours after surgery
  Difference between groups of vasoactive-inotropic score. VIS is calculated as Dopamine dose (mg/kg/min) + Dobutamine dose (mg/kg/min) + 100 x Epinephrine dose (mg/kg/min) + 100 x Norepinephrine dose (mg/kg/min) + 10 x Milrinone dose (mg/kg/min) + 10,000 x Vasopressin dose (units/kg/min).
Neutrophil gelatinase-associated lipocalin concentration | before surgery, immediate ICU admission, 12 and 24 hours after surgery
  Neutrophil gelatinase-associated lipocalin concentrations will be measured in the two groups.
Multiple organ failure | 24 hours after surgery
  Assessment of multiple organ failure through the Sequential organ failure score. The scoring system is mainly divided into 6 parts, namely respiratory function, coagulation function, liver, cardiovascular system, central nervous system, and renal function. The scores range from 0 to 4, with a score of 0 indicating normal function in all organs. The higher the score, the worse the prognosis.
Duration of mechanical ventilation (hours) | 90 days after surgery
  Difference of duration of mechanical ventilation defined as number of hours.
Duration of non-invasive ventilation and High flow oxygen therapy | 90 days after surgery
  Difference of duration of non-invasive ventilation and high flow oxygen therapy defined as number of hours.
ICU stay | 90 days after surgery
  Difference between groups of intensive care unit length of stay defined as number of days.
Hospital stay | 90 days after surgery
  Difference between groups of hospital length of stay defined as number of days.
Major Adverse Kidney Events | 90 days after surgery
  Difference between groups of major adverse kidney events at 90 days after surgery. MAKE is a composite outcome of death, new dialysis and worsened renal function (defined as a 25% or greater decline in eGFR compared to the baseline).
Postoperative pleural and pericardial drainage | 24 hours after surgery
  Difference values between groups of postoperative pleural and pericardial drainage.

OTHER OUTCOMES:
Dose of diuretics and recombinant human brain natriuretic peptide | During CPB surgery, 12 and 24 hours after surgery
  The dosage of diuretics and recombinant human brain natriuretic peptide used during CPB and within 24 hours after surgery will be recorded.
Transfusions | 24 hours after surgery
  Differences between the two groups of transfusions with plasma and stored or autologous red blood cells (RBCs) recovered using intraoperative cell salvage devices.
Renal Ultrasound | immediate admission to ICU, 12 and 24 hours after surgery
  Blood flow grade in renal ultrasound at ICU admission immediately, 12 and 24 hours after surgery
Renal Ultrasound | immediate admission to ICU, 12 and 24 hours after surgery
  Pulsatility index in renal ultrasound at ICU admission immediately, 12 and 24 hours after surgery
Renal Ultrasound | immediate admission to ICU, 12 and 24 hours after surgery
  Resistance index in renal ultrasound at ICU admission immediately, 12 and 24 hours after surgery
Free hemoglobin concentration measure | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Blood free hemoglobin concentrations will be measured in the two groups.
methemoglobin concentration measure | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Blood methemoglobin concentrations will be measured in the two groups.
Nitric oxide metabolite concentration measure | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  The two groups will measure the concentration of nitric oxide metabolites: nitrite (NO2-) and the total of NO metabolites (NOt).
Oxygenation index | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Difference between groups in oxygenation index.
Near-renal infrared oxygen saturation | immediate admission to ICU, 12 and 24 hours after surgery
  Difference between groups in near-renal infrared oxygen saturation.
CVP | before surgery, end of surgery, immediate admission to ICU, 8, 12, 24 hours after surgery
  Differences in values (mmHg) between the two groups of CVP .
PEEP | before surgery, end of surgery, immediate admission to ICU, 8, 12, 24 hours after surgery
  Differences in values （cmH2O） between the two groups of PEEP.
Inflammation related indicators | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Levels of inflammation-related indicators, including the neutrophil lymphocyte ratio(NLR), and the platelet lymphocyte ratio(PLR), will be measured in the two groups.
Inflammation related indicators | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Levels of inflammation-related indicators, including the systemic inflammatory response index(SIRI), and the systemic immune response index(SII) will be measured in the two groups.
Inflammation related indicators | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Levels of inflammation-related indicators, including white blood cell (WBC) will be measured in the two groups.
Oxidative stress related indicators | before surgery, immediate admission to ICU, 12 and 24 hours after surgery
  Levels of oxidative stress-related indicators, including Malondialdehyde (MDA) and superoxide dismutase (SOD) will be measured in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, ICF
Time Frame: Proposals may be submitted up to 6 months following publication of the results of the trial.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.

REFERENCES:
- [Derived] Chen Z, Han X, Li L, Liu M, Yu L, Cheng S, Yu Y, Liu N. Nitric oxide for the prevention of postoperative acute kidney injury in patients undergoing surgery for Stanford type A aortic dissection: study protocol for a randomized controlled trial. Trials. 2025 Aug 11;26(1):284. doi: 10.1186/s13063-025-08986-5. PMID 40790609